CLINICAL TRIAL: NCT01526421
Title: A Randomized Clinical Trial Evaluating the Role of Contingent Reinforcement in the Engagement of and Retention of Drug Users in HAART Programs - Part 1
Brief Title: Use of Incentives to Engage Drug Users in HIV Therapy
Acronym: Incentives-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H11-00592; H11-00592 (Other: UBC/Providence Health Care REB); 1R01DA031043-01 (NIH)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infection
Keywords: HIV; Antiretroviral therapy, highly active
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- monetary reinforcer (Experimental)
  Interventions: Other: monetary reinforcer
- no reinforcer (No Intervention)

INTERVENTIONS:
Other: monetary reinforcer — Participants randomized to the reinforcer arm will receive gift cards at the completion of screening procedures.
  Other Names: contingency management
  Arms: monetary reinforcer

SUMMARY:
Highly active antiretroviral therapy (HAART), the current standard of care for treatment of HIV infection, is highly effective when taken appropriately. Before starting this treatment, a person must be aware of their HIV status and present to a clinic for medical care. They then undergo screening procedures (medical assessment and laboratory tests) to determine whether they are eligible to receive HAART, i.e. whether HIV treatment is necessary and safe for them.

In many urban centres including Vancouver's Downtown Eastside, there is a high rate of HIV infection among users of illicit drugs. However, HIV-infected drug users often do not present to the medical system and complete the process necessary to start HAART. Given the known benefits of HAART, new strategies are required to increase rates of HAART initiation in this group. Contingency management (CM) is a strategy to affect behaviour by providing a reward (e.g. money) to reinforce the desired behaviour. CM has been used with success in other areas of medicine (e.g. smoking cessation, weight loss) and in the drug using population, but has not been established as a means to improve HAART uptake.

The proposed research primarily seeks to assess the effectiveness of monetary-based CM in engaging HIV-infected drug users in HAART programs. Drug users identified through outreach will be randomized in a 1:1 ratio to one of two arms; participants in one arm will be offered a monetary-based reinforcer to participate (n=150) and participants in the second arm will be offered no reinforcer (n=150). Participation involves reporting to the study site for formal study of eligibility screening, consisting of clinical evaluation, medical history and laboratory testing required to determine eligibility to receive HAART. Participants randomized to the reinforcer arm will receive gift cards at the completion of screening procedures.

Our hypothesis is that drug users offered a monetary-based reinforcer will be significantly more likely to complete HAART eligibility screening than those not offered a reinforcer.

DETAILED DESCRIPTION:
HAART eligibility screening entails presenting to the study site within 2 weeks of pre-screening, undergoing laboratory testing and providing a medical history, and returning for results within the subsequent four weeks. Any potential subjects who appear to be acutely intoxicated will be asked to return the next day or at a later date or time of their choosing. All participants will be asked to return for their results within four weeks after screening. Subjects will have 70 mL of whole blood collected by venipuncture by a trained study nurse. Laboratory tests will include HIV confirmatory testing (antibody and Western blot), CD4 cell count and plasma HIV-1-RNA level (plasma viral load; pVL), Hepatitis A, B and C serology, pregnancy test for women of child-bearing potential, complete blood count (CBC) with differential and platelet count, chemistry profile (creatinine, urea and electrolytes), and transaminase levels (ALT, AST). All participants will also have a medical history taken and undergo a physical examination. Recorded data will include subject gender, age, ethnicity, race, area of residence and living arrangement (categorized as homeless/on the street, unstable [defined as living primarily in a single room occupancy hotel, boarding room, or transition house] or stable). Additional features which will be recorded will include nature and frequency of illicit substance use, and participation in other cohort studies or methadone maintenance programs. All clinical past medical history and co-morbidities and laboratory data will be recorded for assessment of subject HAART eligibility.

All subjects who return for the results, whether HAART-eligible or not, will have their laboratory results explained to them and will be counseled as to a recommended course of clinical care by the study nurse. Those eligible for HAART will be offered enrollment into Part II of the study. Those not eligible for HAART will be invited to re-evaluate their eligibility for antiretroviral therapy at yearly intervals through the study site. Once 150 subjects have been randomized to each of the two study arms (total n=300), recruitment will be temporarily halted and statistical analysis will determine whether the reinforcer resulted in a significant and clinically relevant increase in the proportion of subjects who complete HAART eligibility screening.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Self-reports as having used illicit drugs within last 3 months
3. Self-reports known or at-risk for HIV infection.

Exclusion Criteria:

1. Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of interview
2. Has lived in the greater Vancouver area for three months or less (as a means to enhance participant retention)
3. Pregnancy
4. Receipt of antiretroviral therapy within the last 12 months
5. Known history of gambling addiction.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
the proportion of drug users undertaking clinical and laboratory screening to determine eligibility for highly active antiretroviral therapy (HAART). | 6 weeks
  HAART eligibility screening entails presenting to the study site within 2 weeks of pre-screening, undergoing laboratory testing and providing a medical history, and returning for results within the subsequent four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hull, MD, Principal Investigator — University of British Columbia; Julio SG Montaner, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, VIDUS study office site, 342 East Hastings, Vancouver, British Columbia, Canada